CLINICAL TRIAL: NCT04704531
Title: Phase II Clinical Study to Evaluate the Efficacy of Multidose Lagricel® Ofteno Ophthalmic Solution Applied in Three Different Dosage Schemes as Treatment for Mild to Moderate Dry Eye
Brief Title: Phase II Clinical Study to Evaluate the Efficacy of Multidose Lagricel® Ofteno Ophthalmic Solution as Treatment for Dry Eye Disease.
Acronym: PRO-037
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOPH037-1219/II
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — BID protein, human

STUDY DESIGN:
Intervention Model Description: Comparative, controlled, multicenter, open, randomized clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Application of one drop of Multidose Lagricel® Ofteno (Sodium Hyaluronate 0.4%) BID in OU during 30 days.
  Interventions: Drug: Sodium Hyaluronate Ophthalmic 0.4% BID
- Group 2 (Experimental): Application of one drop of Multidose Lagricel® Ofteno (Sodium Hyaluronate 0.4%) QID in OU during 30 days.
  Interventions: Drug: Sodium Hyaluronate Ophthalmic 0.4% QID
- Group 3 (Experimental): Application of one drop of Multidose Lagricel® Ofteno (Sodium Hyaluronate 0.4%) 6 times per day in OU during 30 days.
  Interventions: Drug: Sodium Hyaluronate Ophthalmic 0.4% Six times per day

INTERVENTIONS:
Drug: Sodium Hyaluronate Ophthalmic 0.4% BID — Topical ophthalmic administration of one drop of Multidose Lagricel® Ofteno BID.
  Other Names: PRO-037; Lagricel® Ofteno
  Arms: Group 1
Drug: Sodium Hyaluronate Ophthalmic 0.4% QID — Topical ophthalmic administration of one drop of Multidose Lagricel® Ofteno QID.
  Other Names: PRO-037; Lagricel® Ofteno
  Arms: Group 2
Drug: Sodium Hyaluronate Ophthalmic 0.4% Six times per day — Topical ophthalmic administration of one drop of Multidose Lagricel® Ofteno six times per day.
  Other Names: PRO-037; Lagricel® Ofteno
  Arms: Group 3

SUMMARY:
Phase II, comparative, controlled, multicenter, parallel group, open, randomized clinical study. The main outcome variable will be the Ocular Surface Disease Index (OSDI) questionnaire. Three dosage schemes of topical ophthalmic application of Multidose Lagricel® Ofteno (Sodium Hyaluronate 0.4%; preservative free) are to be evaluated in patients diagnosed with mild to severe dry eye. Each group will be exposed to one of the following administration schemes: 1 drop bis in die (BID), 1 drop quater in die (QID), or 1 drop six times per day; instillation will take place in both eyes (OU).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Being capable of voluntarily grant a signed informed consent.
* Being willing and able to meet the requirements of the study such as attending programmed visits, treatment plan and other study procedures.
* Women in child-bearing age must assure the continuation (start ≥ 30 days prior to informed consent signing) of a hormonal contraceptive method or intrauterine device (IUD) during the study.
* Presenting a mild to moderate dry eye disease diagnosis, defined as:

  * OSDI score between 13 and 32, plus one of the following:

    * More than 5 dots of corneal staining
    * More than 9 dots of conjunctival staining
    * BUT < 10 seconds

Exclusion Criteria:

* Pregnancy, breastfeeding or planning to become pregnant during the time of the study
* Having participated in clinical trials within 30 days prior to signing this study's informed consent form.
* Having participated previously in this study.
* BCVA equal or worse than 20/200, in either eye.
* Diagnosis of any of the following:

  * Allergic, viral or bacterial conjunctivitis
  * Anterior blepharitis
  * Parasite infestation of ocular structures (Demodex, for example)
  * Unresolved history of ocular trauma
  * Scarring diseases of the ocular surface
  * Corneal or conjunctival ulcers
  * Filamentary keratitis
  * Neurotrophic keratitis
  * Bullous keratopathy
  * Neoplastic diseases of the ocular surface or ocular annexes
  * Diseases presenting fibrovascular proliferations on the corneal or conjunctival surface.
  * Any retinal or posterior segment diseases that require treatment or threat the visual outcome.
  * Glaucoma
* Requiring management for dry eye that includes implementation of treatments described in the step 2 management recommendations of the Tear Film & Ocular Surface Society's Dry Eye Work Shop II (TFO DEWS II).
* Previous history of drug addiction within the last 2 years prior to signing this study's informed consent form.
* Having a previous history of any ophthalmological surgical procedure, within the last 3 months prior to the informed consent signing date.
* Being a contact lens user, rigid or soft. Inclusion is possible if the use of contact lenses is suspended both during the study period and at least 15 days prior inclusion takes place.
* Previous history of any medical affliction, acute or chronic, that according to the investigator may increase either the risk to the patient for participating in this study or the risk of interference of the accurate interpretation of results.
* Known hypersensitivity to any of the components of the products used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) | Days: 0 (baseline visit) and 31 (+1) (final visit),
  It is a 12-item questionnaire used to evaluate symptoms associated with dry eye disease, as well as classify their severity. According the obtained score, categories are as follows: normal (0-12 points), mild (13-22 points), moderate (23-32 points), or severe (33-100 points).
Incidence of adverse events | Day 33 (+ 1) (safety call).
  Presence/absence adverse events, defined as the appearance of any unfavorable reaction in a patient participating in a clinical investigation in which any pharmaceutical product is being administered, regardless of the causal attribution.

SECONDARY OUTCOMES:
Change in tear break-up time (BUT) | Days: 0 (baseline visit),15 (± 1) (first follow-up visit), and 31 (+ 1) (final visit).
  After application of fluorescein stain, using a slit lamp and its cobalt blue filter, the time elapsed after instructing the patient to blink 1 or 2 times and the appearance of dry spots on the ocular surface will be counted and reported as BUT. Normally, this parameter is ≥ 10 seconds.
Change in conjunctival and corneal staining with lissamine green | Days: 0 (baseline visit),15 (± 1) (first follow-up visit), and 31 (+ 1) (final visit).
  The evaluation will take place after applying the lissamine green stain on the ocular surface and evaluating the resulting staining pattern. This will be measured through the Oxford scale which includes 6 grades: Absent (0), Minimal (I), Mild (II), Moderate (III), Marked (IV), Severe (V).
Change in conjunctival and corneal staining with fluorescein | Days: 0 (baseline visit),15 (± 1) (first follow-up visit), and 31 (+ 1) (final visit).
  The evaluation will take place after applying the fluorescein stain on the ocular surface and evaluating the resulting staining pattern. This will be measured through the Oxford scale which includes 6 grades: Absent (0), Minimal (I), Mild (II), Moderate (III), Marked (IV), Severe (V).
Change in conjunctival hyperemia | Days: 0 (baseline visit),15 (± 1) (first follow-up visit), and 31 (+ 1) (final visit).
  Rate of conjunctival hyperemia will be evaluated through the Efron scale which includes 5 grades: Normal (0), Very Mild (I), Mild (II), Moderate (3), and Severe (4).
Change in incidence of chemosis | Days: 0 (baseline visit),15 (± 1) (first follow-up visit), and 31 (+ 1) (final visit).
  Chemosis will be evaluated as present (if conjunctiva separates from the sclera in ≥ 1/3 of the palpebral opening area or if it exceeds the eyelid's gray line) or absent.
Change in Best Corrected Visual Acuity (BCVA) | Days: 0 (baseline visit),15 (± 1) (first follow-up visit), and 31 (+ 1) (final visit).
  With the patient's best possible refractive correction, visual acuity will be evaluated through the Snellen chart. Its notation (fraction or decimal) is described as the distance from the chart at which the test is performed, divided by the distance at which a letter equals vertically 5 minutes of arc.
Change in intraocular Pressure (IOP) | Days: 0 (baseline visit),15 (± 1) (first follow-up visit), and 31 (+ 1) (final visit).
  Measured through Goldman tonometer in milligrams of mercury (mmHg). After instillation of topical anesthetic (tetracaine 0.5%) and fluorescein stain, IOP will be evaluated. Normal values are considered between 10 and 21 mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Jalisciense del Metabolismo, S.C., Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No